CLINICAL TRIAL: NCT04135664
Title: Adjuvant Esophagectomy Versus Chemoradiation for Patients With Clinical Stage N0 and Pathological Stage T1b (After Endoscopic Submucosal Dissection, ESD) Esophageal Squamous Cell Carcinoma (Ad-ESD Trial): a Multicentric, Open Label, Randomized Trial
Brief Title: Comparison of Esophagectomy and Chemoradiation for Patients With cN0-pT1b Stage Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Chief of Department of Esophageal Surgery, Deputy of Department of Thoracic Surgery, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chest201908
Record Dates: First submitted 2019-10-09; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Cancer
Keywords: esophagectomy; chemoradiation; esophageal cancer; endoscopic submucosal dissection
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy; Chemoradiotherapy; Watchful Waiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients undergoing adjuvant esophagectomy (Active Comparator): Patients underwent endoscopic submucosal dissection and diagnosed with pathological-T1b and clinical-N0 squamous cell carcinoma.
  Patients randomized into undergoing adjvant esophagectomy.
  Interventions: Procedure: esophagectomy
- Patients undergoing adjuvant chemoradiation (Experimental): Patients underwent endoscopic submucosal dissection and diagnosed with pathological-T1b and clinical-N0 squamous cell carcinoma.
  Patients randomized into undergoing adjvant chemoradiation.
  Interventions: Combination Product: chemoradiation
- Prospective registry of patients that cannot be randomized (Active Comparator): Patients underwent endoscopic submucosal dissection and diagnosed with pathological-T1b and clinical-N0 squamous cell carcinoma.
  Patients cannot be randomized into undergoing adjvant esophagectomy or chemoradiaton.
  This arm includes patients undergoing adjuvant esophagectomy; adjuvant chemoradiation and active surveillance.
  Interventions: Procedure: esophagectomy; Combination Product: chemoradiation; Other: active surveillance

INTERVENTIONS:
Procedure: esophagectomy — esophagectomy with at least two-field (thoracic-abdominal) lymphadenectomy
  Arms: Patients undergoing adjuvant esophagectomy; Prospective registry of patients that cannot be randomized
Combination Product: chemoradiation — concurrent chemotherapy and radiotherapy
  Arms: Patients undergoing adjuvant chemoradiation; Prospective registry of patients that cannot be randomized
Other: active surveillance — No further adjuvant therapy
  Arms: Prospective registry of patients that cannot be randomized

SUMMARY:
The ad-ESD trial is phase III randomized trial to compare adjuvant esophagectomy and chemoradiation for patients with clinical stage N0 and pathological stage T1b squamous cell carcinoma (after endoscopic submucosal dissection).

DETAILED DESCRIPTION:
Esophagectomy is still the primary treatment for pathological T1b esophageal squamous cell carcinoma. However, esophagectomy is associated with high mortality and morbidity and decreased quality of life. Endoscopic resection followed with chemoradiation had showed uncompromised oncological outcomes with esophagectomy. But there is no well-designed, phase III trial to compare the two treatment for patients with pT1b squamous cell carcinoma.

The ad-ESD trial is a multi-center prospective superiority trial, combied of a randomized clinical trial and a prospective registry.

The experimental design produces two randomized arms; (1) esophagectomy and (2) chemoradiation. An additional registry arm will be based on surgeons/patients that do not want to be randomised because of their own experience on adjuvant therapy, including esophagectomy; chemoradiation and active surveillance.

The primary endpoint is to evaluate the difference of 5-year overall survival rate between definitive chemoradiation and esophagectomy, in patients with cN0-pT1b esophageal squamous cell cancer (ESCC) after endoscopic resection.

The secondary endpoints are to evaluate the difference of quality of life and oncological outcomes including 3-year overall survival (OS) and 3, 5-year relapse free survival (RFS) between the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven with esophageal squamous cell cancer.
* Clinical N0 stage diagnosed by imaging examinations.
* Pathological T1b stage confirmed by endoscopic submucosal dissection.
* Age: 18-75.
* Tumor located at the thorax.
* Performance status Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Written informed consent.

Exclusion Criteria:

* Prior intervention treatment before endoscopic submucosal resection.
* Inability to accept any treatment component.
* Prior intervention (surgery, chemoradiation, et al.) for other primary tumor disease.
* Distant metastasis.
* The circumference of the lumen over 3/4
* Main tumor size > 5cm assessed by endoscopy
* Inability to understand the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival rate | 5 years after enrollment day
  The overall survival is defined as days from date of randomization to death from any cause, and cencored at the last day of follow up when patients are alive.

SECONDARY OUTCOMES:
3-year overall survival rate | 3 years after enrollment day
  The overall survival is defined as days from date of randomization to death from any cause, and cencored at the last day of follow up when patients are alive.
3-year relapse free survival rate | 3 years after enrollment day
  The relapse free survival is defined as days from date of randomization until the date of tumor progression or the date of death causing of any reasons, and cencored at the last day of follow up when patients are alive.
5-year relapse free survival rate | 5 years after enrollment day
  The relapse free survival is defined as days from date of randomization until the date of tumor progression or the date of death causing of any reasons, and cencored at the last day of follow up when patients are alive.
Quality of life differences (EORTC QLQ-C30) | 1st, 3rd, 6th, 12th and 24th month after enrollment
  The quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer patients (EORTC QLQ-C30) questionnaire. Patients will be invited to finish the questionnaire at the day of recruitment, 1st, 3rd, 6th, 12th and 24th month after randomization.
Quality of life differences (EORTC QLQ-OES18) | 1st, 3rd, 6th, 12th and 24th month after enrollment
  The quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer patients (EORTC QLQ-OES18) questionnaire. Patients will be invited to finish the questionnaire at the day of recruitment, 1st, 3rd, 6th, 12th and 24th month after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Li, MD, PhD, Principal Investigator — Shanghai Chest Hospital of Shanghai Jiao Tong University
Locations (6):
- China (6):
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Changhai Hospital, The Second Military Medical University, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin

REFERENCES:
- [Derived] Al-Batran SE, Koch C. Neoadjuvant therapy for oesophageal cancer: refining the armamentarium. Lancet. 2024 Jul 6;404(10447):5-7. doi: 10.1016/S0140-6736(24)01084-5. Epub 2024 Jun 11. No abstract available. PMID 38876135
- [Derived] Yang Y, Su Y, Zhang X, Liu J, Zhang H, Li B, Hua R, Tan L, Chen H, Li Z. Esophagectomy versus definitive chemoradiotherapy for patients with clinical stage N0 and pathological stage T1b esophageal squamous cell carcinoma after endoscopic submucosal dissection: study protocol for a multicenter randomized controlled trial (Ad-ESD Trial). Trials. 2020 Jul 1;21(1):603. doi: 10.1186/s13063-020-04461-5. PMID 32611448